CLINICAL TRIAL: NCT03759782
Title: Use of Immune Modulatory Properties of Ribavirin to Enhance Hepatitis B Virus Nucleotide Analog Antiviral Activity: Proposal for Pilot Clinical Trial
Brief Title: Ribavirin to Enhance Hepatitis B Virus Nucleotide Analog Antiviral Activity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180733
Record Dates: First submitted 2018-10-02; First posted 2018-11-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Ribavirin; Tenofovir

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Tenofovir (TDF) 300 mg po once a day (OD)
  Interventions: Drug: Tenofovir
- Group 2 (Active Comparator): Tenofovir 300 mg po OD + Ribavirin 400 mg twice a day (BID) if <70kg / 600 mg every (q) in the morning (AM) and 400 mg q in the evening (PM) if ≥70kg
  Interventions: Drug: Ribavirin; Drug: Tenofovir

INTERVENTIONS:
Drug: Ribavirin — Ribavirin will be added to the standard of care treatment (tenofovir) regime for 24 weeks.
  Arms: Group 2
Drug: Tenofovir — Tenofovir as per standard of care

SUMMARY:
Hepatitis B virus (HBV) leads to life-threatening disease like liver failure and liver cancer. For most, a cure is unattainable as current HBV antiviral therapy (using nucleoside analogues) are not able to clear the virus from their liver. While HBV treatments are typically administered alone (monotherapy), this study will explore the use of Ribavirin in combination with standard therapy to enhance current treatment regimens. Ribavirin is commonly used to treat Hepatitis C Virus (HCV) but there is evidence that Ribavirin also induces immune effects that are beneficial in HBV treatment. The aim of this study is to determine whether combination of Ribavirin and a nucleoside analog is more effective compared to nucleoside analog treatment alone. Enrolled patients will be followed for treatment response according to standard clinical and virological tests, as well as immune response to HBV. Our ultimate goal is to find a more effective treatment and improve health outcomes for persons living with HBV.

ELIGIBILITY:
Inclusion Criteria:

1. HBV Hepatitis B surface antigen (HBsAg) positive for a minimum of 24 weeks
2. HBV DNA level >20,000 IU/mL
3. ≥ 18 years of age

Exclusion Criteria:

1. Willingness and ability to sign an informed consent
2. HBV nucleos(t)ides and/or interferon exposure within 24 weeks of study medication dosing
3. HIV and other immune compromising condition (e.g. cancer with the exception of non-invasive cutaneous malignancy, autoimmune condition) or therapy (i.e. systemic steroids, chemotherapy)
4. HCV co-infected
5. Cirrhosis (defined by biopsy criteria or as >18.4 kilopascal (kPa) by transient elastography)
6. Creatinine Clearance <60 ml/min
7. Baseline hemoglobin <130 g/L in males and <120 g/L in females
8. Unwilling or unable to use contraception (unless confirmed surgical sterilization)
9. Pregnancy confirmed by blood test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The Decline of Participants Serum HBV DNA values for both study arms at each study. | 24 weeks
  The absolute decline in HBV DNA and quantitative HBsAg titre will be compared with baseline level at each study visit overall and between study arms (with or without RBV).

SECONDARY OUTCOMES:
Fibroscan score | 24 weeks
  Individual fibroscan scores pre and post treatment for each group, using fibrosis scores calculated in kilopascal F0 representing no fibrosis and F4 value indicating cirrhosis.
Liver enzyme values | 24 weeks
  Participants individual reduction in liver enzymes at each visit.
Number of participants with treatment related adverse events as assessed by CTCAE v4.0. | 28 weeks
  Safety profile of TDF plus Ribavirin regime

CONTACTS AND LOCATIONS:
Overall Officials: Curtis L Cooper, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - Cumming School of Medicine, University of Calgary, Calgary, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario

REFERENCES:
- [Derived] Keeshan A, Coffin C, Vachon A, Patel N, Fung S, Mortimer L, Crawley A, Ma M, Osiowy C, Cooper C. Ribavirin Does Not Enhance Hepatitis B Virus Nucleotide Antiviral Activity: A Pilot Study. Clin Invest Med. 2022 Dec 31;45(4):E11-15. doi: 10.25011/cim.v45i4.39274. PMID 36586101